CLINICAL TRIAL: NCT04989972
Title: Randomized Double Blind Placebo Controlled Assessing the Efficacy of Micro-dosed Psilocybin in Reducing Anxiety and or Depression Levels in Adults
Brief Title: Assessing the Efficacy of Micro-dosed Psilocybin on Reducing Anxiety & Depression Levels in Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: GCP VIOLATIONS FROM THE SPONSORS
Sponsor: Wake Network, Inc. (Network)
Collaborators: Professor Roger Gibson Section of Psychiatry Faculty of Medical Sciences UWI (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECP242-19/20
Record Dates: First submitted 2021-07-12; First posted 2021-08-04 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2021-06

CONDITIONS: Anxiety and Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — pleurotolysin B, oyster mushroom

STUDY DESIGN:
Intervention Model Description: The research design has a parallel design for the first 8 weeks and a open label single group study for the last 8 weeks
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm (Experimental): participants will take the active intervention PSIL428
  Interventions: Drug: PSIL428
- placebo arm (Experimental): participants will take the intervention 1 mg Oyster mushrooms
  Interventions: Dietary Supplement: Oyster mushroom
- open label (Experimental): all participants will take the active intervention PSIL428
  Interventions: Drug: PSIL428

INTERVENTIONS:
Drug: PSIL428 — 1 mg of psilocybin
  Arms: Intervention arm
Dietary Supplement: Oyster mushroom — 1 mg of oyster mushroom
  Arms: placebo arm
Drug: PSIL428 — 1 mg psilocybin
  Arms: open label

SUMMARY:
To investigate the efficacy of a 16 week treatment with PSIL428 patient reported anxiety levels in otherwise healthy individuals suffering from depression and or anxiety symptoms.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled study assessing the efficacy of micro-dosed psilocybin on reducing anxiety and/or depression levels in adults

Study summary:

The Institute for Health Metrics and Evaluation reported that Anxiety disorders currently affect an estimated 275 million people worldwide, about one in 13 people (7.3 percent).

COVID-19 has accelerated the rate of new anxiety diagnoses and exacerbated pre-existing diagnoses of anxiety in individuals worldwide.

The effectiveness of full dose psilocybin for treatment of anxiety and depression has been shown in a number of clinical trials. While there is a significant evidence of clinical efficacy of full dose psilocybin, acute effects of the dose result in a significant impairment - perceptual and sensory distortions incapacitating the patient for the duration of drug activity. Recent work suggests while not producing perceptual changes, micro-dosing may indeed be associated with improved mood and enhanced well-being. The practice of micro-dosing is gaining popularity in the general population, while clinical data on its safety and efficacy is lacking.

This will be a novel randomized, double-blind, placebo-controlled study aimed at establishment of safety and anxiolytic efficacy of psilocybin PSIL428 administered in a micro-dosing regimen (2-5% of a full therapeutic dose) to adults suffering from depression or anxiety.

The primary outcome of this study is the change in anxiety and/or depression levels from screening to week 16. Participant anxiety levels will be monitored through Beck Anxiety inventory, depression levels - through Beck Depression Inventory forms on a bi-weekly basis across the course of the study.

Study Drug PSIL428 is an experimental intervention and the active ingredient psilocybin is botanically derived. Similar interventions are currently undergoing Phase IIb/III clinical trials in international jurisdictions. It is being assessed for treatment of depressive disorders. Typically psilocybin used in full therapeutic doses associated with significant acute adverse effects. The proposed trial would utilize psilocybin in different dosing regimen - as micro-dosing - ingesting of sub-perceptual doses of the drug equal to 2-10% of the full dose. The micro-dosing practice is gaining significant popularity world-wide, however evidence-based data around it is minimal. Risks and benefits associated with the trial are not definitively established, however existing pre-clinical and clinical data around full-dose use of the drug carries a favorable risk-benefit potential.

The trial will be conducted in accordance with the most recently acceptable version of the Declaration of Helsinki, Good Clinical Practice (GCP) according to International Conference on Harmonization (ICH) guidelines, and applicable Standard Operating Procedures (SOPs). The trial will be conducted under a protocol reviewed and approved by an IRB; the trial will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the subjects will be respected; each subject will give his or her written informed consent before any protocol-driven tests or evaluations are performed.

The investigators are responsible for obtaining informed consent in adherence to GCP and according to applicable regulations prior to entering the subject into the trial.

A positive change in Beck Anxiety and/or Beck Depression numeric levels between PSIL428 and placebo groups will mark our primary outcome achievement of confirming beneficial effects of micro-dose-administered psilocybin on study participants' overall anxiety and/or depression levels

ELIGIBILITY:
Inclusion Criteria:

* Experiencing persistent anxiety and/or depression symptoms
* Scoring between 10-20 on BAI and/or between 15-25 on BDI-II
* Females and males with the minimum age of 18 at screening;
* Not of child bearing potential, which is defined as females who have had hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with 1 year since last menstruation)

OR

* Female participants of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result, prior to enrollment. All hormonal birth controls require a minimum stability of three months and remain consistent throughout the study. Acceptable methods of birth control include:
* Hormonal contraceptives; oral, hormone patch (Ortho Evra), vaginal ring (NuvaRing), injectable (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method
* Intrauterine devices
* Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
* Vasectomy of partner (shown successful as per appropriate follow-up);
* Willing to maintain current levels of activity throughout the study;
* Healthy as determined by self-report and medical history;
* Willingness to complete all study visits and requirements associated with the study;
* Has access to a computer, tablet, or smart phone with internet connection; sufficiently comfortable with using app-based technology for data gathering;
* Has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria

* Individuals who are pregnant, breastfeeding, or planning to become pregnant.
* Individuals with psychotic disorders including schizophrenia; bipolar disorder. personality disorder. Participants with 1st-degree relatives with related psychotic disorders.
* Alcohol or drug abuse within the last 6 months that meets the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria.
* Participation in a clinical research study within 30 days of enrollment.
* Allergy or sensitivity to study product ingredients.
* Clinically significant abnormal laboratory results at screening.
* Unstable medical conditions as assessed by the Principal Investigator.
* Individuals who are cognitively impaired and/or unable to give informed consent.
* Any other condition which in the Principal Investigator's opinion may adversely affect the participant's ability to complete the study or its measures or which may pose significant risk to the participant.
* Individuals who have taken a psychedelic drug (Psilocybin, DMT, Peyote, Ayahuasca, Ibogaine, LSD, Ketamine) within 60 days of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Beck Anxiety Inventory BAI | Screening to week 16
  Measures 21 items in physical and cognitive anxiety ranges 0-7 mild, to 26-63 severe
  Questionnaire BDI-11
Changes in Beck Depression Inventory 02 - BDI-II | screening to week 16
  Measures 21 items in the presence and severity of depressive symptoms 0-9 no depression, 10 -18 mild depression, 19-29 moderate to severe depression

SECONDARY OUTCOMES:
Change in the European Quality of life 5 dimensions- EQ-5D | screening to week 16
  changes between the intervention PSIL-428 and placebo groups for mobility, self-care, pain & discomfort, usual activities and anxiety & depression
Cognitive flexibility, using the Stroop Color & Word Test (SCWT) | Screening to week 16
  Changes in cognition between the PSIL-428 and placebo groups in the reading of words as compared to identifying & naming colors. A stopwatch is used and the test-taker reads color words or names ink colors from different pages as quickly as possible. An interference score, cognitive flexibility, creativity and reaction to cognitive pressure are measured
Changes in resilience using the Brief Resiliency Scale | Screening to 16 weeks
  assesses the ability of the individual to bounce back or recover from stress a score of one means low resiliency and a score of 5 means high resiliency
Measurement of higher level cognitive processes using the Wisconsin Card Sorting Test | screen to 16 weeks
  Uses two card packs, having 4 stimulus cards and 64 response cards measures attention, perseverance , abstract thinking and set shifting.
The incidence of adverse events | Screening to 16 weeks
  The number of reported cases of adverse events
The severity of adverse events | Screening to 16 weeks
  Adverse events which range from mild,moderate, severe and lethal
Incidence of abnormal blood pressure | Screening to 16 weeks
  Blood pressure which is consistently above and below120/80
Incidence of abnormal heart rate | Screening to 16 weeks
  The incidence of atrial fibrillation, supraventricular tachycardia or bradycardia
incidence of irregular heart rate | Screening to 16 weeks
  incidence of arrhythmias
incidence of suicidal ideation using the Columbian Suicide Severity Rating Scale | Screening to 16 weeks
  Measures Suicidal Ideation items 1-5; Suicidal Behavior 6-10 and both Suicidal Ideation and Behavior Items 1-10
Change in the number of steps | Screening to Week 16
  Wearable and or mobile devices
Changes in concomitant medication | Screening to 16 weeks
  Recently prescribed medication
Changes in volume of Alcohol | screening to 16 weeks
  self reports
Changes in the number of cigarettes | screening to 16 weeks
  self reports
Changes in the number of cannabis joints | Screening to 16 weeks
  Self reports
Changes in other over the counter medication | Screening to 16 weeks
  Self Reports
Changes in Estradiol | Screening to 16 weeks
  Salivary panel profile values
Changes in Testosterone | Screening to 16 weeks
  Salivary panel profile vales
Changes in Cortisol | Screening to 16 weeks
  Salivary panel profile values
Changes in Progesterone | Screening to 16 weeks
  Salivary panel profiles values
Changes in Melatonin | Screening to 16 weeks
  Salivary panel profile values
Changes in DHEA (Dehydroepiandrosterone) | Screening to 16 weeks
  Salivary panel profile values
Changes in DHT(Dihydrotestosterone) | Screening to 16 weeks
  Salivary panel profile values
Changes in Androstenedione | Screening to 16 weeks
  Salivary panel profile values
Changes in Estrone | Screening to 16 weeks
  Salivary panel profile values

CONTACTS AND LOCATIONS:
Overall Officials: Roger Gibson, Principal Investigator — Faculty of Medical Sciences UWI Mona; Sharon White, Study Director — Wake Network, Inc.
Locations (1):
- FMS Department of Psychiatry, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: No
The data will be made available through publications and conference presentations